CLINICAL TRIAL: NCT02256618
Title: A Pilot Feasibility and Safety Study of Autologous Umbilical Cord Blood Cell Therapy in Infants With Neonatal Encephalopathy
Brief Title: Autologous Cord Blood Cell Therapy for Neonatal Encephalopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neonatal Encephalopathy Consortium, Japan (Network)
Collaborators: Osaka City University (Other); Yodogawa Christian Hospital (Other); Kurashiki Central Hospital (Other); Nagoya University (Other); Osaka City General Hospital (Other); Saitama Medical University (Other); National Cerebral and Cardiovascular Center, Japan (Other); National Center for Child Health and Development, Japan (Unknown); Tokyo University (Other); Tokyo Women's Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMIN000014903
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Neonatal Encephalopathy; Hypoxic-ischemic Encephalopathy
Keywords: neonatal encephalopathy; hypoxic-ischemic encephalopathy; newborn infants; neonates; umbilical cord blood cells
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cell therapy (Experimental): Infants who are born at the study sites, have moderate to severe encephalopathy, and have cord blood available for infusion
  Interventions: Other: Autologous umbilical cord blood cells

INTERVENTIONS:
Other: Autologous umbilical cord blood cells — Autologous non-cryopreserved volume- and red blood cell-reduced cord blood cells will be intravenously infused

SUMMARY:
This is a pilot study to test feasibility and safety of intravenous infusion of autologous umbilical cord blood cells in the first 72 hours after birth if a neonate is born with signs of encephalopathy.

DETAILED DESCRIPTION:
This is a multicenter pilot study to evaluate the feasibility and safety of intravenous infusions of autologous (the patient's own) umbilical cord blood cells in term gestation newborns with neonatal encephalopathy (hypoxic-ischemic encephalopathy). If a neonate is born with signs of moderate to severe encephalopathy and cooled for the encephalopathy, the neonate can receive their own non-cryopreserved volume- and red blood cell-reduced cord blood cells. The cord blood cells are divided into 3 doses and infused at 12-24, 36-48, and 60-72 hours after the birth. Infants will be followed for safety and neurodevelopmental outcome up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

Infants are eligible if they meet all the following inclusion criteria except 4.

1. ≥36 weeks gestation
2. Either a 10-minute Apgar score ≤5, continued need for resuscitation for at least 10 minutes, or severe acidosis, defined as pH <7.0 or base deficit ≥16 mmol/L in a sample of umbilical cord blood or any blood during the first hour after birth
3. Moderate to severe encephalopathy (Sarnat II to III)
4. A moderately or severely abnormal background amplitude-integrated EEG (aEEG) voltage, or seizures identified by aEEG, if monitored
5. Up to 24 hours of age
6. Autologous umbilical cord blood available to infuse within 3 days after birth
7. A person with parental authority must have consented for the study.

Exclusion Criteria:

1. Known major congenital anomalies, such as chromosomal anomalies, heart diseases
2. Major intracranial hemorrhage identified by brain ultrasonography or computed tomography
3. Severe growth restriction, with birth-weight less than 1800 g
4. Severe infectious disease, such as sepsis
5. Hyperkalemia
6. Outborn infants (Infants born at hospitals other than the study sites)
7. Volume of collected cord blood <40 ml
8. Infants judged critically ill and unlikely to benefit from neonatal intensive care by the attending neonatologist

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2014-08; Primary Completion 2017-10 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Adverse event rates | first 30 postnatal days
  Adverse event rates (combined rate of death, continuous respiratory support, and continuous use of vasopressor) will be compared between the cell recipients and historical controls at 30 days of age.

SECONDARY OUTCOMES:
Efficacy | 18 months
  Neuroimaging at 12 months of age and neurodevelopmental function at 18 months of age will be compared between the cell recipients and historical controls.

CONTACTS AND LOCATIONS:
Overall Officials: Haruo Shintaku, MD, PhD, Study Director — Osaka City University
Locations (6):
- Japan (6):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Saitama Medical University, Kawagoe, Saitama
  - Yodogawa Christian Hospital, Osaka
  - Osaka City General Hospital, Osaka
  - Osaka City University, Osaka

REFERENCES:
- [Background] Tsuji M, Taguchi A, Ohshima M, Kasahara Y, Sato Y, Tsuda H, Otani K, Yamahara K, Ihara M, Harada-Shiba M, Ikeda T, Matsuyama T. Effects of intravenous administration of umbilical cord blood CD34(+) cells in a mouse model of neonatal stroke. Neuroscience. 2014 Mar 28;263:148-58. doi: 10.1016/j.neuroscience.2014.01.018. Epub 2014 Jan 18. PMID 24444827
- [Background] Ohshima M, Taguchi A, Tsuda H, Sato Y, Yamahara K, Harada-Shiba M, Miyazato M, Ikeda T, Iida H, Tsuji M. Intraperitoneal and intravenous deliveries are not comparable in terms of drug efficacy and cell distribution in neonatal mice with hypoxia-ischemia. Brain Dev. 2015 Apr;37(4):376-86. doi: 10.1016/j.braindev.2014.06.010. Epub 2014 Jul 14. PMID 25034178
- [Background] Taguchi A, Soma T, Tanaka H, Kanda T, Nishimura H, Yoshikawa H, Tsukamoto Y, Iso H, Fujimori Y, Stern DM, Naritomi H, Matsuyama T. Administration of CD34+ cells after stroke enhances neurogenesis via angiogenesis in a mouse model. J Clin Invest. 2004 Aug;114(3):330-8. doi: 10.1172/JCI20622. PMID 15286799